CLINICAL TRIAL: NCT06502925
Title: Evaluation of the Quality of Incoming Call Handling Assisted by the proQA Software in the Emergency Dispatch Center of Besançon.
Brief Title: Quality of Incoming Call Handling in an Emergency Dispatch Center
Acronym: CRRAQPA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/833
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Medical Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of Emergency Medical Dispatch (EMD) is to ensure prompt access to medical care for all at all times, initiate appropriate responses quickly, arrange suitable hospital facilities, and coordinate patient transport and hospitalization.

In France, care begins with an incoming call managed by the EM Dispatchers, who collect the patient's details and assess the seriousness of the situation. This severity assessment is essential for triggering the appropriate resources: direct dispatch of first-aiders in extreme emergencies, or transfer of the call to an emergency or general practitioner.

Under- or over-assessment will necessitate redirection, resulting in a loss of time and opportunity for the patient, or emergency channel congestion. Errors at this stage can impact the entire care pathway.

To assist EM dispatchers, aids have been developed. Firstly, In France, a diploma course was created in 2019. Various training methods exist. Their contribution to the quality of incoming calls handling remains unevaluated. Secondly, EM centers use regulation protocols designed to guide dispatchers in call handling and identifying the seriousness of the situation.

The regulation protocol used at Besançon University Hospital is ProQA (Priority Dispatch Corporation, Salt Lake City, UT, US). It uses standardized questions and records EM Dispatchers' decisions and the responses they obtain from callers. These responses are considered by ProQA, which then assigns a "severity" code to the call.

The assistance provided by regulation protocols, however useful, remains insufficient. Contextual factors can complicate compliance with regulation protocols, making matching resources to needs challenging.

AQUA is a software package dedicated to quality control, enabling EM Dispatcher's supervisors to rate the quality of all stages of the call-taking process. This ensures that all key questions have been asked and that they have been asked correctly. In addition, the 'severity' code obtained by the EM Dispatcher can be compared with the 'severity' code obtained by the supervisor, using a qualifying analysis method and data entry software. The calls are replayed under optimal conditions, in a calm environment and allowing supervisors to listen multiple times to ensure no information is missed. the supervisors' code is therefore the reference code.

CRRAQPA study's aim is to assess the quality of incoming call handling and to identify the factors that influence this quality.

ELIGIBILITY:
Inclusion Criteria:

* Calls handled by a professional EM Dispatcher during the study period.

Exclusion Criteria:

* Calls handled by a medical student functioning as an EM Dispatcher.
* Calls for which the "severity" code is unfounded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will study incoming calls in the EMD of Besançon University Hospital. These calls must be handled by a professional EM dispatcher and must have a 'severity' code that is not unfounded.
  During the replay and evaluation, it can happen that the supervisor is unable to assign a severity code with certainty. This occurs when a decisive question regarding the severity code has not been asked, and the information has not been provided spontaneously by the caller. In such cases, the supervisor considers the code obtained by the EMD to be unfounded
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of incoming calls for which the 'severity' code identified by the EM dispatchers during the call and the 'severity' code identified by the supervisor after replaying the call are in agreement. | Through study completion, the anticipated duration is 1 year
  The quality of the incoming call will be assessed based on the agreement between the 'severity' code identified by the EM dispatchers during the call and the 'severity' code identified by the supervisor after replaying the call using the AQUA software.
  There are six possible severity codes, which will be grouped into a three-category variables corresponding to the three possible referrals (emergency physician, general practitioner, 'flash' departure).

SECONDARY OUTCOMES:
The proportion of over- and under-rated calls. | Through study completion, the anticipated duration is 1 year
  An over-rated call occurs when the severity level identified by the EM dispatcher is higher than that identified by the supervisor upon replay.
  An under-rated call occurs when the severity level identified by the EM dispatcher is lower than that identified by the supervisor upon replay
The proportion of the different training modalities received by EM dispatchers. | Through study completion, the anticipated duration is 1 year
  In France, several training modalities exist for EM dispatchers such as field training, 2019 diploma training, training via tape replay, call simulation training.
The number of years of experience in the profession of the EM dispatchers participating in the study. | Through study completion, the anticipated duration is 1 year
The rate of answered calls within 20 s (= quality of service at 20 seconds, QS20) | Through study completion, the anticipated duration is 1 year
The number of calls per hour in the call centre. | Through study completion, the anticipated duration is 1 year
The duration between the beginning of the EM dispatcher's shift and the time at which the incoming call occurs | Through study completion, the anticipated duration is 1 year
The proportion of incoming calls occurring during the day or night | Through study completion, the anticipated duration is 1 year
The proportion of incoming call occuring during week days or week-ends | Through study completion, the anticipated duration is 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Leclerc, Principal Investigator — University Hospital of Besançon
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besancon, Besançon, Franche Comté
  - University Hospital of Besançon, Besançon, Franche Comté

IPD SHARING:
Plan to Share IPD: Yes
The data in this study are not publicly available, but reasonable requests can be made.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date
Access Criteria: Researchers who submit a methodologically sound proposal approved by our research team